CLINICAL TRIAL: NCT05763303
Title: Impact of an Interventional Program on Self-Management Among Students With Diabetes in Assiut University
Brief Title: Impact of an Interventional Program on Self-Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ramadan Ali Hamza, Physician at The Health Directorate in Asyut Governorate, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Diabetes Self Management
Record Dates: First submitted 2023-02-10; First posted 2023-03-10 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Self Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): received interventional program which will consist of :
  1. -The educational part: the health education intervention will be in the form of brief counselling five sessions (about half an hour for each session at 1-week intervals) which are introduced after data collection and blood analysis by simplified manner, in the study's clinic.
  2. Training part: We will invite every participant to join this part of the program which will be performed in the fitness center of the faculty of physical education, Assiut University. The entire duration of the 8-week exercise training program is closely supervised by 2 qualified personnel. The exercise session includes running or walking on treadmill, and cycling on bicycle ergometer, about 30 minutes, 3 times per week,
  Interventions: Other: educational program
- control group (Other): traditional care: the participants will received traditional care in health facility but nothing by researcher
  Interventions: Other: educational program

INTERVENTIONS:
Other: educational program — interventional program consists of educational part and training part in case of agreement of participants

SUMMARY:
The goal of this randomized clinical trial study is to assess the effect of an interventional program on diabetes self-management and therefore on effective glycemic control among diabetic students in Assuit university

DETAILED DESCRIPTION:
1. To formulate a strategy aiming to reduce the burden of diabetes morbidity & mortality;
2. To determine degree of self-management in diabetic participants
3. To identify the obstacles facing the diabetic students to achieve an accepted self-management;
4. To assess the impact of the interventional program on overcoming such obstacles; and
5. To assess the impact of diabetes self-management on glycemic control among diabetic students in Assiut University All university students who suffer from diabetes and attend the study's clinic seeking medical treatment during a full academic year (2023/2024) with inclusion and exclusion criteria are recruited. The sample is divided into 150 cases for intervention group and 150 for control group (traditional care), by Systemic random technique. All participants will be exposed to Questionnaires for assessment of Diabetes Self-management, and measurements of glycated hemoglobin (HbA1c), body weight, height, at base line, three months, and 6 months after the end of the program.

ELIGIBILITY:
Inclusion Criteria:

•Confirmed cases of diabetes mellitus (IDD" type I" & NIDD "type II") among Assiut University students

Exclusion Criteria:

* Diabetic students with severe disability or handicapped
* Diabetic students known to have another health problem make him un tolerable to do exercise such as cardiovascular disease, bronchial asthma
* Diabetic students with speech and hearing difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
assessment of change in Perceived Obstacles to diabetes self-management that faced by participants | at base line, three months and six months after the end of the program.
  by short version of the diabetic obstacle questionnaire.
assessment of Change in Diabetes Self-management | at base line, three months and six months after the end of the program.
  by diabetes self-management questionnaire,
assessment of change in measurements of glycated hemoglobin (HbA1c) | at base line, three months and six months after the end of the program.
  by blood analysis to measure (HbA1c)

SECONDARY OUTCOMES:
assessment of change in measurement of body mass index (BMI) | at base line, three months and six months after the end of the program.
  by measurement of weight in kilograms and height in meters and use formula: (BMI) = weight in kilograms ÷ ( height in meter × height in meter)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hassan Qayed, Chair, Study Chair — Assiut University; Manal El-Sayed EzzEl-Dine Abdel-Mooty, director, Study Director — Internal Medicine - Assiut faculty of Medicine; Emad Shaban Ali Hassan, director, Study Director — Department of Sports Health Sciences, Faculty of Physical Education
Locations (1):
- faculty of medicine / Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No